CLINICAL TRIAL: NCT02631694
Title: Targeting Fear Memory by Disrupting the Process of Reconsolidating: A New Intervention for Panic Disorder
Brief Title: Disruption of Memory Reconsolidating as a Treatment for Panic Disorder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Mrs. M. Kindt, Professor of Experimental and Clinical Psychology, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MKAEWC1
Record Dates: First submitted 2015-12-09; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Propranolol; Carbon Dioxide; Compressed Air

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (3):
- Fear reactivation with propranolol (Experimental)
  Interventions: Drug: Propranolol; Other: Carbon dioxide
- Fear reactivation with placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Other: Carbon dioxide
- No fear reactivation with propranolol (Placebo Comparator)
  Interventions: Drug: Propranolol; Other: Compressed air

INTERVENTIONS:
Drug: Propranolol — Intake of propranolol pill (40 milligram)
  Arms: Fear reactivation with propranolol; No fear reactivation with propranolol
Drug: Placebo — Intake of placebo pill (40 milligram)
  Arms: Fear reactivation with placebo
Other: Carbon dioxide — Inhalation of 35% carbon dioxide
  Arms: Fear reactivation with placebo; Fear reactivation with propranolol
Other: Compressed air — Inhalation of air
  Arms: No fear reactivation with propranolol

SUMMARY:
Animal and human fear conditioning studies have repeatedly shown that administering propranolol before or after retrieval of a previously acquired fear results in an elimination of the fear expression. This approach, known as disruption of fear memory reconsolidation, is a promising new avenue for treating anxiety disorders. The present study aims to test its efficacy in patients with panic disorder.

ELIGIBILITY:
Inclusion Criteria:

* a primary diagnosis of panic disorder according to DSM-V
* written approval of an independent physician for participation

Exclusion Criteria:

* other relevant treatment for panic disorder at the time of study - e.g., Cognitive Behavioral Therapy (CBT)
* diagnosis of depression
* diagnosis of psychosis
* use of psychotropic medication
* history of pulmonary diseases
* metabolic acidosis
* history of cardiovascular diseases
* heart problems among first-degree relatives
* heart rate (HR) < 60
* blood pressure (BP) < 90-60 or BP > 170-100
* history of black-outs or fainting
* diabetes
* liver or kidney diseases
* hyperactive production of thyroid hormones
* epilepsy
* any medication contra-indicative of the use of propranolol
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change in the number of participants diagnosed with panic disorder assessed by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, fourth addition (DSM-IV) Axis I Disorders | Baseline and 3 months
Change in score on the Panic Disorder Severity Scale (PDSS-SR) | Baseline, 7 days, 3 months

SECONDARY OUTCOMES:
Carbon dioxide challenge using a visual analogue scale ranging from 0-100 mm | 3 months
  Participants are asked to rate on a visual analogue scale ranging from 0-100 mm the degree to which they are willing to inhale carbon dioxide again if this were requested. Secondly, participants will indeed be requested to perform the challenge a second time and rate on the visual analogue scale how anxious it made them feel.
Change in score on the Panic Appraisal Inventory (PAI) | Baseline, 7 days, 3 months, 6 months, 1 year
Change in score on the Mobility Inventory (MI) | Baseline, 7 days, 3 months, 6 months, 1 year
Change in score on the Body Sensations Questionnaire (BSQ) | Baseline, 7 days, 3 months, 6 months, 1 year
Change in score on the Agoraphobic Cognitions Questionnaire (ACQ) | Baseline, 7 days, 3 months, 6 months, 1 year
Change in the number of participants diagnosed with panic disorder assessed by the Structured Clinical Interview for DSM-IV Axis I Disorders | Baseline, 6 months, 1 year
Change in score on the Panic Disorder Severity Scale (PDSS-SR) | Baseline, 6 months, 1 year

OTHER OUTCOMES:
Score on the Anxiety Sensitivity Index (ASI) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Merel Kindt, Prof. dr., Principal Investigator — University of Amsterdam